CLINICAL TRIAL: NCT02190305
Title: Rapid Diagnostics for HIV and Hepatitis - Multiplo HBc/HIV/HCV and Reveal HBsAg
Brief Title: Rapid Diagnostics for HIV and Hepatitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: MedMira Laboratories Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCP002
Record Dates: First submitted 2014-07-09; First posted 2014-07-15 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: HIV Infections; Hepatitis B Infections; Hepatitis C Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic: Multiplo HBc/HIV/HCV + Reveal HBsAg (Experimental): Subjects tested with investigational devices and approved comparator assay algorithms for HIV and hepatitis B and C.
  Interventions: Device: Multiplo HBc/HIV/HCV and Reveal HBsAg

INTERVENTIONS:
Device: Multiplo HBc/HIV/HCV and Reveal HBsAg — All subjects tested with both investigational devices, plus with algorithms of approved assays for HIV and hepatitis B and C.
  Other Names: Multiplo Rapid HBc/HIV/HCV Antibody Test; Reveal Rapid Hepatitis B Surface Antigen Test

SUMMARY:
The purpose of this study is to determine the efficacy of two rapid diagnostic tests in plasma, venipuncture whole blood, and fingerstick whole blood. The clinical performance of Multiplo HBc/HIV/HCV will be determined by comparing the results with patient infected status for HIV-1/2 (human immunodeficiency viruses 1 and 2), HBV (hepatitis B virus) and HCV (hepatitis C virus). The clinical performance of Reveal HBsAg will be determined by comparing the results with patient infected status for HBV.

Subject participation in the study will consist of a single one-hour visit, at which time blood samples will be drawn for testing with the investigational devices and with approved comparator assays. The test results, which are the outcome of the study, will be obtained only once, at the time of this visit.

DETAILED DESCRIPTION:
The objective of this study is to determine the performance characteristics of two rapid diagnostic tests.

Approximately 3000-4500 subjects in total will be enrolled in the study into four different study populations. In Population 1, which is "at risk" group of about 2000-3000 subjects, roughly 2/3 will be individuals who are at risk of infection with HIV or hepatitis B or C, or who have signs or symptoms of hepatitis. Approximately 500 of these individuals are expected to be known HIV-positive individuals.

The remaining three study populations will be comprised of individuals with known infection with HIV (Population 1A, ~500 individuals), HBV (Population 1B, ~500 individuals), and HCV (Population 1C, ~500 individuals).

Both Multiplo HBc/HIV/HCV and Reveal HBsAg will be used to test finger stick whole blood, venous whole blood and plasma samples from each subject in Population 1. Plasma samples (repository or fresh) will be used to fulfill the requirements for Populations 1A, 1B, and 1C.

For all enrolled subjects, the plasma sample will be tested with the following FDA-approved assays: EIA for anti-HIV-1/2, anti-HCV, anti-HBc total, anti-HBc IgM, anti-HBs, and HBsAg. The efficacy of Multiplo will be determined by comparing the results with patient infected status for HIV-1/2, HBV and HCV. The efficacy of Reveal will be determined by comparing the results with patient infected status for HBV.

The primary analysis will involve comparison of Multiplo HBc/HIV/HCV and Reveal HBsAg results for each of the test markers (anti-HIV-1/2, anti-HCV, anti-HBc, and HBsAg), in each sample matrix (finger stick whole blood, venous whole blood and plasma) with the patient infected status as determined by separate algorithms for HIV, HBV, and HCV. The percent positive and percent negative agreement will be determined relative to patient infected status for each marker and sample type, with corresponding two-sided 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* 13 years of age or older
* able to sign consent form (or parent/guardian sign consent plus subject sign assent for ages 13-18)
* willing to complete the risk assessment questionnaire, and
* willing to provide blood samples: finger stick sample (2 drops), 1 serum separator tube, 2 anticoagulant (K2 EDTA) tubes.

Population 1 - Diagnostic Trial "At Risk" Group (n = 2000-3000)

Subjects must meet one or more of the following inclusion criteria to be enrolled in Population 1:

* Have at least one risk factor for infection with hepatitis B or C,
* Have at least one risk factor for infection with HIV,
* Present with signs and symptoms of hepatitis,
* Be a known HIV-positive individual (previous positive HIV test result, may comprise up to 500 individuals)

Population 1A - Additional known HIV-positive individuals (n = ~500)

Subjects must:

• be a known HIV-positive individual (previous positive HIV test result).

Population 1B - Additional known HBV-positive individuals (n = ~500)

Subjects must:

• be known to have current or past HBV infection, as evidenced by HBV serology results.

Population 1C - Additional known HCV-positive individuals (n = ~500)

Subjects must:

• be known to be infected with HCV, as evidenced by previous positive HCV test results.

Exclusion Criteria:

* Subjects do not meet the inclusion criteria

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05 (Estimated); Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of Reveal HBsAg and Multiplo HBc/HIV/HCV | At single study visit
  For each enrolled subject, Multiplo HBc/HIV/HCV and Reveal HBsAg devices will be used to test finger stick whole blood, venipuncture whole blood, and plasma samples. Plasma will also be tested using separate algorithms of FDA approved assays to determine patient infected status for HIV-1/2, hepatitis B, and hepatitis C.
  The performance of Reveal HBsAg will be determined relative to patient infected status for hepatitis B for each matrix assessed. The performance of Multiplo HBc/HIV/HCV will be determined relative to patient infected status for each of hepatitis B, HIV-1/2, and hepatitis C.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Schiff, MD, Principal Investigator — University of Miami; Peter Kerndt, MD, Principal Investigator — University of Southern California - Los Angeles; Fabienne Laraque, MD, Principal Investigator — New York City Department of Health and Mental Hygiene
Locations (4):
- United States (4):
  - Keck School of Medicine - LAUSC, Los Angeles, California
  - SCFLD Hepatology Diagnostic Research Laboratory, Miami, Florida
  - Minneapolis Medical Research Foundation, Minneapolis, Minnesota
  - NYC Dept Health & Mental Hygiene, New York, New York